CLINICAL TRIAL: NCT05974540
Title: Ultrasound Versus Physical Examination for Cricothyroid Membrane Determination in Pediatric Patients
Brief Title: USG vs Palpation for Cricothyroid Membrane Determination
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof., Marmara University
Other Study IDs: 09.2023.605
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-08

CONDITIONS: Ultrasound; Cricothyroid Membrane
Keywords: Cricothyrotomy; Palpation; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Determination of cricothyroid membrane — After the patient's head is extended, the pediatric surgeon will be asked to mark the cricothyroid membrane with a pencil using traditional inspection and palpation methods. Then, the cricothyroid membrane will be determined by the Anesthesiology and Reanimation specialist by USG method and the difference will be determined. Demographic and morphometric characteristics of the patients will be recorded. In addition, the length of the cricothyroid membrane, the distance between the cricoid cartilage and the skin, the distance between the cricoid cartilage and the 2nd tracheal ring will be measured by USG.
  Mallampati classes of patients with intubation, Cormack-Lehane (CL) glottic appearance grades, Likert scale with intubation difficulties (1: very easy, 2: easy, 3: medium, 4: difficult) will also be recorded.

SUMMARY:
Emergency cricothyroidotomy is a very important technique to ensure airway safety in acute situations. Problem in identifying the cricothyroid membrane is a major contributor to high failure, as the most common complication during cricothyrotomy is the misplacement of the cannula. The success rate of emergency airway access performed by anesthesiologists and emergency medicine specialists was found to be low due to the low frequency of the procedure. The aim in this study is to compare the palpation method with the ultrasonugraphy (USG)-based method in determining the cricothyroid membrane. The hypothesis is that USG is more successful than palpation in identifying the cricothyroid membrane. In addition, the relationship between difficult intubation and measurements such as the cricothyroid membrane length, the cricoid cartilage and the skin distance, the distance between the cricoid cartilage and the second tracheal ring will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) I and II physical status
* Elective pediatric surgery
* Patients going to be intubated

Exclusion Criteria:

* ASA III or above physical status
* Emergency surgery
* Patients having tracheostomy
* Patients going to have laryngeal mask

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients between the ages of 1-18, who are in ASA I-II physical status and who will undergo elective surgery under general anesthesia by the Pediatric Surgery at Marmara University Pendik Training and Research Hospital will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Distance between palpation-based and USG-based determination of the cricothyroid membrane | On the 1 day of the surgery. After the anesthesia induction and intubation.
  Regarding the determination point of the cricothyroid membrane the distance between palpation-based method performed by pediatric surgeon and USG-based method performed by anesthesiologist will be measured.

SECONDARY OUTCOMES:
Cricothyroid membrane length | On the 1 day of the surgery. After the anesthesia induction and intubation.
  Cricothyroid membrane length will be measured by anesthesiologist using USG. Longitudinal view of the thyroid, cricoid and trakeal ring cartilages will be obtained and the measurement will be made.
Skin distance from cricoid cartilage | On the 1 day of the surgery. After the anesthesia induction and intubation.
  Skin distance from cricoid cartilage will be measured by anesthesiologist using USG. Longitudinal view of the thyroid, cricoid and trakeal ring cartilages will be obtained and the measurement will be made.
Distance between cricoid cartilage and 2nd tracheal ring | On the 1 day of the surgery. After the anesthesia induction and intubation.
  Distance between cricoid cartilage and 2nd tracheal ring will be measured by anesthesiologist using USG. Longitudinal view of the thyroid, cricoid and trakeal ring cartilages will be obtained and the measurement will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Ruslan Abdullayev, Principal Investigator — Marmara University Department of Anesthesiology and Reanimation
Locations (1):
- Marmara University Department of Anesthesiology and Reanimation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided